CLINICAL TRIAL: NCT05618561
Title: EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test Clinical Performance Study
Brief Title: EuGeni Rapid Antigen Test for the Qualitative Detection of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Causing COVID19 Disease in Compliance With the World Health Organization (WHO)
Acronym: WHO
Status: Terminated | Type: Observational
Why Stopped: High number of false negatives
Sponsor: AnteoTech Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CT013
Record Dates: First submitted 2022-11-10; First posted 2022-11-16 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: SARS-CoV-2 Infection
Keywords: covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nasopharyngeal specimen collection arm: Specimens collected in nasopharyngeal form from positive subjects with symptoms and negative subjects hospitalized and negative subjects with respiratory symptoms.
  Interventions: Diagnostic Test: EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test
- Combined nasal mid-turbinate and throat specimen collection arm: Specimens collected in combined nasal mid-turbinate form from positive subjects with symptoms and negative subjects hospitalized and negative subjects with respiratory symptoms.
  Interventions: Diagnostic Test: EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test

INTERVENTIONS:
Diagnostic Test: EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test — Subjects have two swabs taken for analysis, one (combined or nasopharyngeal) with the kit under investigation and the other (by standard of care) for analysis with PCRl.

SUMMARY:
Rapid antigen detection (RAD) tests are used to perform rapid diagnosis of SARS-CoV-2 infection based on a qualitative approach. RAD tests detect the viral antigen by the immobilized coated SARS-CoV-2 antibody placed on the device. The results of these tests are available in a short time, reducing the workload in diagnostic hospitals and laboratories and improving the turn-around time.

EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test is an in vitro Diagnostic (IVD) medical device intended to be used for the qualitative detection of SARS-CoV-2 nucleocapsid antigen. The result from this IVD test identifies the presence or absence of the SARS-CoV-2 antigen as an aid for the diagnosis of COVID-19 infection.

DETAILED DESCRIPTION:
The EuGeni SARS-CoV-2 Antigen (Ag) Rapid Detection Test (RDT) is a test strip based on lateral flow technology which utilizes nanoparticles, doped with europium, as the fluorescence reporter system. The test strip is housed in a cassette which is read by the EuGeni AX-2X-S Reader, a portable instrument that reads EuGeni fluorescent lateral flow tests.

The test line contains an immobilized monoclonal mouse antibody to capture SARS-CoV-2 antigen and the control line contains an immobilized control anti-mouse antibody.

The test sample is added to the sample well of the test cassette and then reconstitutes the dried europium nanoparticle antibody conjugate from the conjugate pad. The sample flows along the test strip by capillary action.

If the sample contains SARS-CoV-2 antigen, it binds to the antibody-labelled europium nanoparticle. When the sample flows past the test line, the europium bound antigen is captured by the second anti-SARS-CoV-2 antibody immobilized on the test line. A fluorescent signal detected by the EuGeni AX-2X-S Reader at this test line indicates that the specimen is SARS-CoV-2 antigen Positive.

If the sample does not contain SARS-CoV-2 antigen, the europium-labelled anti-antigen antibody will not bind to the test line. This indicates that the specimen is SARS-CoV-2 antigen Negative.

The sample continues to flow along the strip and when it passes over the control line, antibody-labelled europium nanoparticles are captured by the immobilized anti-mouse antibody. The control line must be detected by the EuGeni AX-2X-S Reader for the test to be valid. If the control line is not detected, the test is considered invalid and must be repeated using another test cassette.

ELIGIBILITY:
Inclusion Criteria:

1. Specimens from subjects over 12 years old agreeing to participate in the study and with a legal representative able to provide informed consent, OR;
2. Specimens from subjects over 18 years old able to provide informed consent.
3. Specimens collected with nasopharyngeal swabs, OR;
4. Combined nasal mid-turbinate and throat specimen collection.

Exclusion Criteria:

1. Specimens and testing methods that are not deemed to be in line with gold-standard RT-PCR standards.
2. Specimens stored for over 2 hours at 2-8 ºC temperature between collection and testing with EuGeni SARS-CoV-2 Ag RDT.
3. Specimens stored for over 5 days at -20ºC between collection and testing with RT-PCR.
4. Specimens stored for over 24h at 4ºC between collection and testing with RT-PCR.
5. Contamination and/or deterioration of the specimen which, in the opinion of the investigator, may affect its handling and/or analysis.
6. The subject is deemed unsuitable to participate in the study by the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The entire population over 12 years of age that met the inclusion criteria and none of the exclusion criteria. Positive subjects must present COVID19 symptoms. In the case of negative subjects, one part must be hospitalized (for any reason) and the other part must have respiratory symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 599 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic sensitivity and specificity in terms of true positive results and true negative results between the kit under investigation and the gold-standard PCR | Through study completion, an average of 4 months
  Number of true positives and true negatives in terms of sensitivity and specificity (accuracy) by contrasting the result obtained with the investigational kit and the gold-standard PCR result.

SECONDARY OUTCOMES:
The sensitivity and the specificity values between the two collection methods, nasal and nasopharyngeal. | Through study completion, an average of 4 months
  To compare the sensitivity and specificity value translated as true positives and true negatives between the investigational kit and PCR between the two sample collection methods, nasal and nasopharyngeal.

CONTACTS AND LOCATIONS:
Overall Officials: M. Antonia Sánchez Calavera, Principal Investigator — C.S. Fuentes Norte
Locations (5):
- Institut Virion, Split, Croatia
- Laiko General Hospital, Athens, Greece
- Spain (3):
  - Centro de Salud Fuentes Norte, Zaragoza, Aragon
  - Centro de Salud Torre Ramona, Zaragoza, Aragon
  - Hospital Universitario de A Coruña (CHUAC), A Coruña, Galicia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/61/NCT05618561/Prot_001.pdf
  • Statistical Analysis Plan (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT05618561/SAP_002.pdf